CLINICAL TRIAL: NCT06427720
Title: Competitive Endogenous Role of the LINC00511/miR-185-3p Axis and miR-301a-3p From Liquid Biopsy as Molecular Markers for Breast Cancer Diagnosis
Brief Title: LINC00511/miR-185-3p Axis and miR-301a-3p Markers for Breast Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Prof. Nadia M. Hamdy, Ph.D., Professor of biochemistry and molecular biology, Ain Shams University
Other Study IDs: RHDIRB2020110301REC#259
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Early Diagnosed Breast Cancer
Keywords: easy diagnosed; stage I/II; Non treated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Four milliliters of peripheral blood was withdrawn once from controls and BC patients, at the time patients were first diagnosed clinically with BC and before any medical (neo)adjuvant therapy or surgical intervention, under strict sterile conditions, following standard biosecurity and international safety procedures, into polymer gel vacutainers with a clot activator (Greiner Bio-One GmbH, Australia), left for 15 min at room temperature to clot, followed by a 10-min centrifugation at 10,000g at 4°C. Sera obtained were aliquoted into three clean Eppendorf tubes and stored at -80°C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: free from any medical, psychosocial, emotional conditions, or cancer (age interval was 28-82) were included in the study as well, matched with BC patients' group in sex and race, menopausal status, and randomly chosen from the female Egyptian population.
- BC patients: full family disease/cancer history was recorded, as well as patients' previous surgical procedures, other than breast surgery, that do not affect the tumor burden, such as splenectomy, tonsillectomy, cesarean birth, and plastic surgery, offspring numbers, menopausal or not, and taking hormonal contraceptives or not.
  Patients' individual current cancer status and the tumor clinical assessment, done at the NCI, using the tumor-node-metastasis (TNM) categorization (43) and the Bloom-Richardson Scale for histological grading (44), were collected from patients' data files, after a biopsy was taken at the time of BC examination

SUMMARY:
Breast cancer is a leading cause of death among women globally, with significant incidence in Egypt. It is characterized by aggressive behavior and resistance to treatment, necessitating early detection methods. Research has revealed that many cancer-related mutations are in non-coding DNA, including microRNAs (miRNAs) and long non-coding RNAs (LncRNAs). miRNAs like miR-185-3p and miR-301a, and LncRNAs such as LINC00511, are potential biomarkers for cancer diagnosis due to their roles in gene regulation and stability in circulation. This study aims to explore the diagnostic utility of these biomarkers in breast cancer.

DETAILED DESCRIPTION:
1. Introduction 1.1. Background: Breast cancer is one of the leading causes of death for women globally, according to the world health organization (WHO), the number of cancer cases expected in 2025 will be 19.3 million cases. In Egypt, cancer is an increasing problem and especially breast cancer [1].

   Breast cancer is the most common female malignant tumor and a major threat to women's health and its development is considerably aggressive local invasion, early metastases, and multidrug resistance to chemotherapy [2, 3]. Therefore, developments of minimally-invasive markers for early detection of breast cancer are of great interest.

   The cancer genome Atlas (TCGA) revealed that many of the mutations and copy number changes found in cancer do not overlap with protein coding genes [4], but are frequently located in non-coding DNA-including non-coding RNA genes [5]. MicroRNAs (miRNAs) were among the first non-coding RNAs to be investigated cancer, and their roles as therapeutic targets or biomarkers in cancer [6].

   MiRNAs are short, single-stranded RNA sequences (usually 19-23 nucleotides) that control gene expression in a variety of physiological and developmental process, thus having a critical role in posttranscriptional regulation of gene expression in a broad range of biological systems [7, 8]. MiRNAs mediate the repression of target mRNA by base pairing to complementary sequence in the 3'-UTR, causing transcript destabilization, translational repression or both [9]. It has been reported that miRNAs also modulate gene expression by binding to other regions, including protein-coding exons [10], and can even induce gene expression in mammalian cells [11].

   Cell-free circulating miRNAs usually exist bound to ribonucleoprotien complexes or high-density lipoprotein or they are released from cells in lipid vesicles, micro-vesicles, exosomes or apoptotic bodies [12-15].Thus, circulating miRNAs may reflect homeostatic response of the organism, as well as signs of disease progression. Owing to their stability and resistance to endogenous RNAse activity, these miRNAs have been proposed as diagnostic and prognostic biomarkers for diseases, including cancer [16].

   Among these miRNAs, MiR-185-3p has been identified as a tumor suppressor gene in various types of cancer. The expression of miR-185-3p was decreased in breast cancer cells MDA-MB-231, and MCF-7. Moreover, miR-185-3p was over-expressed in the LINC00511 silenced transfection, while decreased in the enhancedLINC00511 plasmid transfection [17].

   MicroRNA-301a is another oncomiR that has been related to tumor progression in several types of cancer. For example, in prostate cancer, gastric cancer as well as pancreatic cancer [18-21]. However, its role in breast cancer is not fully investigated.

   Long non-coding RNA (LncRNAs) are those longer than 200 nucleotides, and many of them can also act as primary transcripts to produce short RNAs. Generally, LncRNAs have been implicated in gene-regulatory roles, such as chromatin dosage compensation, imprinting, epigenetic regulation, cell cycle control, nuclear and cytoplasmic trafficking, and cell differentiation [22]. Furthermore, pre-mRNA interaction where the primary transcript is interacting with LncRNAs and ends up with a different functional spliced sequence or is degraded into endogenous small interfering RNAs, miRNA sponges, modulation of protein activity or localization and facilitation of riboprotein complex formation. Not in the least, LncRNAs can stand as precursors for smaller fragments like miRNAs or piRNAs. The main function of ciRNAs consists in miRNAs capturing through complementary interactions, functioning like miRNAs sponge [23]. LncRNAs have already been implicated in human disease including cancer [24].

   Long intergenic noncoding RNA 00511 (LINC00511); is an oncogene that influences tumor size, metastasis, and poor prognosis. LINC00511 binds histone methyltransferase EZH2 and specifies the histone modification pattern on p57 [25]. It also acts as an oncogene in squamous cell carcinoma and pancreatic ductal adenocarcinoma [26]. In particular, little is known whether LncRNAs can serve as biomarkers for cancer prognosis or diagnosis. [27] 1.2. Problem: The role of these biomarkers are not investigated yet in breast cancer early diagnosis.

   1.3. Hypothesis: Tumor Suppressor or Oncogenic Biomarkers and LncRNA used in early diagnosis of breast cancer"
2. Aim of the Work:

   The ultimate aim of the work is to provide a clearer picture of the functions of miR-185-3p, miR-301a, in association with LINC00511in the early diagnosis of breast tumors with measuring both sensitivity and specificity.
3. Previous Studies Findings: in half page. No previous clinical studies were made on the aspect of the diagnostic utilities of the studied biomarkers.
4. Problem Statement:

   The role of these biomarkers are not investigated yet in breast cancer early diagnosis in Egyptian patients.
5. Research Significance:

Primary Outcome:

• To identify Peripheral blood circulating Tumor Suppressor or Oncogenic Small Biomarkers breast cancer and to compare with normal control expression

Secondary Outcome:

• To calculate sensitivity and specificity of miR-185-3p, miR-301a, and LINC00511 as compared to the protein-based markers (CEA and CA15-3) as diagnostic markers.

6. Research Objectives:

1. Analyze the expression level of two miRNA (miR-185-3p, miR-301a) and their predicted interacted lncRNA (LINC00511) as minimal noninvasive molecular markers for diagnosing the primary breast cancer.
2. Compare miR-185-3p, miR-301a, and LINC00511 with the protein based markers (CEA and CA15-3) as diagnostic markers, regarding to sensitivity and specificity.
3. Study the relation between miR-185-3p, miR-301a, and LINC00511and the clinicopathological characters of breast cancer.
4. Research Methodology:

This study will first be approved by the Ethical Committee of Faculty of Pharmacy, Ain Shams University and by the Ethical Committee of National Cancer Institute, New Cairo. Moreover, it will be performed in adherence to the Declaration of Helsinki Guidelines, where two groups will be included and all subjects will give their written consent, to be archived.

Group 1 the control group: A total of 50 healthy volunteers' who are age matched healthy female volunteers not suffering from any disease or taking any medication.

Group 2 (Malignant Breast Tumor): 50 women with non-metastatic primary breast cancer Patients recently diagnosed who haven't yet received any chemotherapy or radiotherapy, attending the National Cancer Institute, New Cairo.

Full history will be taken for all cases and control. The characteristics of the breast cancer patients with regards to age, menopausal status, histopathological type, tumor size, lymph node metastasis and tumor grade, as well as estrogen receptor (ER) and progesterone receptor (PR) will be collected for data analysis.

Exclusion criteria

Patients with:

* Blood disorder diseases, -Any cancer other than breast cancer
* Liver Cirrhosis, Uterine & Urinary bladder diseases

Methods:

Routine Work:

Blood Sampling:

5 ml blood will be collected into plain vaccutainer tubes for serum preparation. Serum samples will be stored at -80 ºC until biochemical assessment at the Biochemistry Department Research Lab, Faculty of Pharmacy, Ain Shams University.

Assay of miR-185-3p, miR-301a, and LINC00511by Quantitative PCR:

MiRNA and LncRNAs will be extracted from serum using Qiagen miRNeasy Mini Kit according to the manufactures' protocol and their concentration and purities will be detected by nanodrop spectrophotometer.

Enriched RNA will be reverse transcribed with miroRNA or LncRNAs reverse transcription kit according to the manufactures' protocol.

Expression of miRNA and LncRNAs will be quantified by qRT-PCR using human MicroRNA and LncRNAs assay kits and their specific primers.

The expression levels of the investigated miRNA will be evaluated using the ∆Ct method [28]. The cycle threshold (Ct) value is the number of qPCR cycles required for the fluorescent signal to cross a specific threshold. ∆Ct will be calculated by subtracting the Ct values of RNU6-2 and GAPDH from those of investigated miRNAs and LncRNAs, respectively. The ∆∆Ct will be calculated by subtracting the ∆Ct of the control samples from the ∆Ct of the cancer samples.

Examination of Hormone Receptors and Protein-based tumor Markers: Both estrogen receptor, progesterone receptor and human epidermal growth factor receptor 2 (HER-2neu), in addition to CEA and CA15.3 tumor markers using ELISA kits will be obtained from National Cancer Institute, New Cairo.

SAMPLE SIZE ESTIMATION The aim of this study is to investigate the Role of some circulating MiRNAs from independent control and breast cancer cases with 1 control per experimental subject. Based on previous study(Hu et al. 2012) the oncogenic small biomarkers expression was normally distributed with standard deviation 2.9 and large effect size (1.09). If the true differences in the breast cancer group and control group means is 2.25 we will need to study 25 experimental subjects and 25 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05.

As regards the tumor suppressor expression means was normally distributed with large effect size (1.4). If the true differences in the breast cancer group and control group means is 14 we will need to study 15 experimental subjects and 15 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05.

Total sample size will be 80 cases, this number will be increased by 25% for expected losses, and total sample is 100 subjects, 50 subjects per group.

Sample size estimation was performed by G power* sample size calculator.

Statistical Analysis:

SPSS 21.0 software package (SPSS,Chicago,IL) will be used to perform the statistical analyses. T-test or Mann-Whitney's U test will be used to compare the difference of continuous variables in two groups as appropriate. Pearson's Chi-square analysis or Fisher's exact test will be employed to compare the difference of categorical variables. Receiver operating characteristic (ROC) curve and area under the ROC curve (AUC) will be plotted to determine the best cutoff point that discriminates between cancer and non-cancer groups; the sensitivities and specificities will be calculated for the miRNAs and their diagnostic efficacy For all analyses, a two-tailed P value of 0.05 or less will be considered as statistically signiﬁcant.

5. Research Time Plan/Frame i. Time plan Q/year Actions Q1 Preparation of the official documents for sample collection, data collection and ethical approval and calculate sample size for control and patients Q2 Sample collection from patients with selected criteria and separation of serum in aliquots Q3 Continue sample collections and separation of serum in aliquots + Extraction of RNA from the samples Q4 Collection of control samples and Extraction of RNA Q1 cDNA synthesis for all samples + qPCR Q2 Statistical analysis of the data and starting to write a paper + collection of related articles for thesis writing Q3 Publication of the paper and finalizing the thesis for revision

ii. Paper title: "The Diagnostic Utility of Tumor Suppressor or Oncogenic Small Biomarkers in Association with LncRNA in Breast Cancer"

Authors:

Marwa M. Mohamed, Dr. Eman Fouad Sanad, Dr. Reham Ali Abbas El-Shimy, Nadia M. Hamdy.

Corresponding Submitting Author: Prof. Nadia M. Hamdy First Author: Marwa M. Mohamed Contributing Author(S): Dr. Eman Fouad Sanad, Dr. Reham Ali Abbas El-Shimy

6. References List:

1. D. A. Ragab, M. Sharkas, S. Marshall, and J. Reen,"Breast cancer detection using deep convolutional neural networks and support vector machines," PeerJ, vol. 7, p. e6201, 2019.
2. A. E. Cyr and J. A.Margenthaler,"Molecular profiling of breast cancer, "Surgical Oncology Clinics of North America, vol. 23, no. 3. Pp. 451-462, 2014.
3. W. J. Gradishar,"Treatment of metastatic breast cancer, "in JNCCN Journal of the National Comprehensive Cancer Network, 2014, vol. 12, no. 5 SUPPL., pp, 759-761.
4. H. L. Martin, L. Smith, and D. C. Tomlinson, "Multidrug-resistant breast cancer: Current perspectives, "Breast Cancer: Targets and Therapy, vol. 6, no. 0. Pp. 1-13, 2014.
5. S. Nik-Zainal et al., "Landscape of somatic mutations in 560 breast cancer whole-genome sequences, "Nature, vol. 534, no. 7605, pp. 47-54, 2016.
6. M. T. Maurano et al., "Systematicc localization of common disease-associated variation in regulatory DNA," Science (80-.)., vol. 337, no. 6099, pp. 1190-1195, 2012.
7. M. V. Iorio and C. M. Croce, "MicroRNA dysregulation in cancer: Diagnostics, monitoring and therapeutics. A comprehensive review, "EMBO Molecular Medicine, vol. 4, no. 3. Pp. 143-159, 2012.
8. D. Baek, J. Villen, C. Shin, F. D. Camargo, S. P. Gygi, and D. P. Bartel, "The impact of microRNAs on protein output, "Nature, vol. 7209, pp. 64-71, 2008.
9. L. P. Lim et al., "Microarray analysis shows that some microRNAs downregulate large numbers of target mRNAs, "Nature, vol. 433, no. 7027, pp. 769-773, 2005.
10. W. Filipowicz, S. N. Bhattacharyya, and N. Sonenberg, "Mechanisms of post-transcriptional regulation by microRNAs: Are the Answers in sight?," Nature Reviews Genetics, vol. 9, no. 2. Pp. 102-114, 2008.
11. J. J. Forman, A. Legesse-Miller, and H. A. Coller,"A search for conserved sequences in coding regions reveals that the let-7 microRNA targets Dicer within its coding sequence, "Proc. Natl. Acad. Sci., vol. 105, no. 39, pp. 14879-14884, 2008.
12. S. Vasudevan, Y. Tong, and J. A. Steitz, "Switching from repression to activation: MicroRNAs can up-regulate translation, "Science (80-.)., vol. 318, no. 5858, pp. 1931-1934, 2007.
13. K. C. Vickers, B. T. Palmisano, B. M. Shoucri, R. D. Shamburek, and A. T. Remaley, "MicroRNAs are transported in plasma and delivered to recipient cells by high-denisty lipoproteins, "Nat. Cell Biol., vol. 13, no. 4, pp. 423-435, 2011.
14. H. Valadi, K. Ekstrom, A. Bossios, M. Sjostrand, J. J. Lee, and J. O. Lotvall, "Exosome-mediated transfer of mRNA and microRNAs is a novel mechanism of genatic exchange between cells., "Nat. Cell Biol., vol. 9, no. 6, pp. 654-9, 2007.
15. J. L. Lindenberg et al., "Funcional delivery of viral miRNAs via exosomes, "Proc. Natl. Acad. Sci., vol. 107, no. 14, pp. 6328-6333, 2010.
16. A. Turchinovich, L. Weiz, and B. Burwinkel, "Extracellular miRNAs: The mystery of their origin and function, "Trends Biochem. Sci., vol. 37, no. 11, pp. 460-465, 2012.
17. L. J. Chin and F. J. Slack, "A truth serum for cancer---- microRNAs have major potential as cancer biomarkers, "Cell Res., vol. 18, no. 10, pp. 983-984, 2008.
18. Lu et al, "Journal of Experimental & Clinical Cancer Research" (2018)
19. Cui, L. et al. Expression of MicroRNA-301a and its Functional Roles in Malignant Melanoma. Cellular physiology and biochemistry: international journal of experimental cellular physiology, biochemistry, and pharmacology 40, 230-244, (2016).
20. Shi, Y. K., Zang, Q. L., Li, G. X., Huang, Y. & Wang, S. Z. Increased expression of microRNA-301a in nonsmall-cell lung cancer and its clinical significance. Journal of cancer research and therapeutics 12, 693-698, (2016).
21. Chen, Z. et al. miR-301a promotes pancreatic cancer cell proliferation by directly inhibiting Bim expression. Journal of cellular biochemistry 113, 3229-3235, (2012).
22. Ma, X. et al. Modulation of tumorigenesis by the pro-inflammatory microRNA miR-301a in mouse models of lung cancer and colorectal cancer. Cell discovery 1, 15005, (2015).
23. O. Wapinski and H. Y. Chang, "Long noncoding RNAs and human disease," Trends in Cell Biology, vol. 21, no.6. pp. 354-361, 2011.
24. D. Gulei, N. Mehterov, S. M. Nabavi, A. G. Atanasov, and I. Berindan-Neagoe, "Targeting ncRNAs by plant secondary metabolites: The ncRNAs game in balance towards malignancy inhibition, "Biotechnology advances, vol. 36, no. 6. Pp. 1779-1799, 2018.
25. T. Derrien, R. Guigo, and R. Johnson, "The long non-coding rnas: A new (p)layer in the 'dark matter, "Frontiers in Genetics, vol. 2, no. Jan. 2012.
26. Ding J, Yang C, Yang S. LINC00511 interacts with miR-765 and modulate tongue squamous cell carcinoma progression by targeting LAMC2. J Oral Pathol Med. 2018;47:46876.
27. Zhao X, Liu Y, Li Z, Zheng S, Wang Z, Li W, Bi Z, Li L, Jiang Y, Luo Y, Lin Q, Fu Z, Rufu C. Linc00511 acts as a competing endogenous RNA to regulate VEGFA expression through sponging hsa-miR-29b-3p in pancreatic ductal adenocarcinoma. J Cell Mol Med. 2018;22:655-67
28. S. H. Kim et al., "Correlation of ultrasound finfings with histology, tumor grade, and biological markers in breast cancer, "ActaOncol. (Madar)., vol. 47, no. 8, pp. 1531-1538, 2008.
29. M. H. Zweig and G. Campbell, "Receiver-operating characteristic (ROC) plots: A fundamental evaluation tool in clinical medicine, "Clinical Chemistry, vol. 39, no. 4. Pp. 561-577, 1993.

(30)Hu, Z. B., J. Dong, L. E. Wang, H. X. Ma, J. B. Liu, Y. Zhao, J. H. Tang, X. Chen, J. C. Dai, Q. Y. Wei, C. Y. Zhang & H. B. Shen (2012) Serum microRNA profiling and breast cancer risk: the use of miR-484/191 as endogenous controls. Carcinogenesis, 33, 828-834.

ELIGIBILITY:
Inclusion Criteria:

* were being an adult female, with breast invasive carcinoma of no specific type, confirmed pathologically

Exclusion Criteria:

* Patients with:
* were blood disease, any cancer other than BC, liver cirrhosis, and uterine and urinary bladder diseases, or metastatic BC patients who received chemo/radiotherapy, or had previous mastectomy.

Ages: 28 Years to 82 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The current retrospective cohort study included 70 female volunteer patients first diagnosed with primary BC, without any medical or surgical intervention, from the Clinical Oncology Department, NCI, Cairo University, Egypt. BC diagnosis is carried out with mammogram and MRI.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
1. Analyze the expression level of two miRNA (miR-185-3p, miR-301a) and their predicted interacted lncRNA (LINC00511) | 12 Month
  as minimal noninvasive molecular markers for diagnosing the primary breast cancer.
2. Compare miR-185-3p, miR-301a, and LINC00511 | 6 Month
  with the protein based markers (CEA and CA15-3) as diagnostic markers, regarding to sensitivity and specificity.
3. Study the relation between miR-185-3p, miR-301a, and LINC00511 | 2 Month
  LINC00511and the clinicopathological characters of breast cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Advanced Biochemistry Research Lab, Cairo, Egypt